CLINICAL TRIAL: NCT05481645
Title: Evaluating the Efficacy and Safety of TQB2450 Injection Combined With Chemotherapy ± Anlotinib Hydrochloride Capsules for First-line Treatment of Patient With Advanced Endometrial Cancer or Sarcoma of Uterus: a Multi-center, Open-label, Randomized Controlled, Phase II Clinical Trial.
Brief Title: Efficacy and Safety of TQB2450 Injection Combined With Chemotherapy ± Anlotinib Hydrochloride Capsules for Advanced Endometrial Cancer or Sarcoma of Uterus.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Per sponsor request. Premature closure was not prompted by any safety or efficacy concerns.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-II-14
Record Dates: First submitted 2022-07-06; First posted 2022-08-01 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Advanced Endometrial Cancer; Sarcoma of Uterus
MeSH Terms: interventions — Carboplatin; Paclitaxel; Doxorubicin; Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group one (Experimental): First-line treatment: TQB2450 injection 1200mg,d1/Q3W+Carboplatin Injection, AUC=5 mg/ml.min,d1/Q3W + Paclitaxel Injection 175mg/m2,d1/Q3W;6-8 cycles;
  Maintenance treatment: TQB2450 injection, 1200mg，d1/Q3W
  Interventions: Drug: TQB2450 injection; Drug: Carboplatin Injection; Drug: Paclitaxel Injection
- Group two (Experimental): First-line treatment: TQB2450 Injection 1200mg, d1/Q3W + Anlotinib Hydrochloride Capsules 8mg/qd, d8-21/Q3W + Carboplatin Injection AUC=5 mg/ml.min, d1/Q3W + Paclitaxel Injection 175mg/m2, d1/Q3W ; 6-8 cycles; Maintenance treatment: TQB2450 injection+ Anlotinib Hydrochloride Capsules 8mg/qd, d8-21/Q3W
  Interventions: Drug: TQB2450 injection; Drug: Anlotinib Hydrochloride Capsule; Drug: Carboplatin Injection; Drug: Paclitaxel Injection
- Group three (Experimental): First-line treatment stage:
  TQB2450 injection 1200mg, d1/Q3W + anlotinib hydrochloride capsules 8mg/qd, d8-21/Q3W+ chemotherapy（① Doxorubicin Hydrochloride Injection 60mg/㎡，d1/Q3W; or ② Gemcitabine Hydrochloride Injection 900mg/㎡, d1, d8/Q3W+ Docetaxel Injection 75mg/㎡, d8/Q3W）; 6-8 cycles;
  Maintenance phase:
  TQB2450 injection 1200mg, d1/Q3W+ Anlotinib hydrochloride capsules 10mg/qd, d8-21/Q3W
  Interventions: Drug: TQB2450 injection; Drug: Anlotinib Hydrochloride Capsule; Drug: Doxorubicin Hydrochloride Injection; Drug: Gemcitabine Hydrochloride Injection; Drug: Docetaxel injection

INTERVENTIONS:
Drug: TQB2450 injection — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents the binding of PD-L1 to PD-1 and B7.1 receptors on the surface of T cells, thereby reactivating T cells and enhancing the immune response.
Drug: Anlotinib Hydrochloride Capsule — Anlotinib hydrochloride is a muti-target tyrosine kinase inhibitor.
  Arms: Group three; Group two
Drug: Carboplatin Injection — Carboplatin which s similar to alkylating agent, is a second-generation platinum anti-tumor drug, which mainly causes cross-linking of DNA within and between chains, destroys DNA molecules, and disintegrates the helix.
  Arms: Group one; Group two
Drug: Paclitaxel Injection — Paclitaxel is a diterpene alkaloid with anticancer activity
  Arms: Group one; Group two
Drug: Doxorubicin Hydrochloride Injection — Doxorubicin hydrochloride is a cycle non-specific anticancer chemotherapy drug, which directly acts on DNA, changes the nature of DNA template, and inhibits DNA polymerase.
  Arms: Group three
Drug: Gemcitabine Hydrochloride Injection — Gemcitabine is a cell cycle specific antimetabolic drug, which mainly acts on tumor cells at the DNA synthesis stage.
  Arms: Group three
Drug: Docetaxel injection — Docetaxel is an anti-tumor drug of paclitaxel, which plays an anti-tumor role by interfering with the microtubule network necessary for cell Mitosis and interphase cell function.
  Arms: Group three

SUMMARY:
This clinical study plans to enroll 69 endometrial cancer patients and 5-10 uterine sarcoma patients. The trial is divided into a lead-in phase and a main phase. The lead-in phase will include 9 subjects, while the main phase will enroll 60 endometrial cancer patients randomized 1:1. Additionally, 5-10 uterine sarcoma patients will be enrolled. The study aims to evaluate the efficacy and safety of TQB2450 injection combined with chemotherapy ± anlotinib hydrochloride capsules as first-line treatment, followed by TQB2450 injection monotherapy ± anlotinib hydrochloride capsules as maintenance therapy for advanced endometrial cancer or uterine sarcoma. The study will also explore efficacy-related biomarkers, mechanisms of action, safety and/or pathological mechanisms, and surgical conversion rates. The primary endpoint is ORR (Objective Response Rate).

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily participated in this study, signed the informed consent, and had good compliance;
* Age: ≥18 years old (when signing the informed consent form); ECOG PS score: 0-1; expected survival period of more than 3 months; body mass index (BMI) > 18.5 and weight > 40kg;
* Who have not received first-line systemic anticancer therapy and are not suitable for receiving treatment other than systemic treatment:

  1. Group 1 and 2: Stage III/IV epithelial endometrial cancer (including endometrioid carcinoma, non-endometrioid carcinoma, carcinosarcoma) confirmed by histopathology, and the subject also needs to meet one of the following categories:

     1. Newly diagnosed subjects: there are still residual lesions visible on imaging after non-radical surgery;
     2. Subjects with initial recurrence: if the subject received systemic platinum-based adjuvant and/or neoadjuvant chemotherapy，and the recurrence time is more than 6 months from the end of the last chemotherapy，then the previous chemotherapy is allowed.
  2. Group 3: Stage I-IV sarcoma of uterus, and the subject also needs to meet one of the following categories:

     1. Newly diagnosed/initial recurrence subject of high grade endometrial stromal sarcoma (ESS)、undifferentiated Uterine sarcoma (UUS) , uterine Leiomyosarcoma and adenosarcoma(uLMS) with sarcoma overgrowth (OS). The definition of new diagnosis and initial recurrence is the same as above.
     2. Low grade ESS, adenosarcoma without SO and other Uterine sarcoma with ER+/PR+，the subjects who failed in antiestrogen treatment.
* According to the RECIST 1.1 criteria, there is at least one measurable lesion. If the measurable lesion is located in the area of previous radiotherapy, it should be clearly defined as progressing state;
* Tumor tissue samples can be provided to detect MSI/MMR status or traceable test reports;
* The main organs function well and meet the following standards:

  1. Blood routine examination standards (no blood transfusion within 7 days before screening, no correction with hematopoietic stimulating factor drugs):

     1. Hemoglobin (HGB) ≥90 g/L;
     2. The absolute value of neutrophils (NEUT)≥1.5×109/L;
     3. Platelet count (PLT) ≥ 90 × 109/L;
  2. The biochemical examination shall meet the following standards:

     1. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN);
     2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN. If accompanied by liver metastasis, ALT and AST≤5×ULN;
     3. Serum creatinine (Cr) ≤ 1.5×ULN or creatinine clearance (Ccr) ≥ 60ml/min;
     4. Serum albumin (ALB)>30g/L;
  3. Urine routine examination standard: urine routine indicates urine protein <++; if urine protein ≥++, it is necessary to confirm the 24-hour urine protein quantitative ≤1.0g;
  4. Coagulation function or thyroid function tests should meet the following criteria:

     1. Prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (INR) ≤ 1.5×ULN (no anticoagulation therapy);
     2. Thyroid-stimulating hormone (TSH) ≤ ULN; T3 and T4 levels should be investigated if abnormal, and normal T3 and T4 levels can be selected.
  5. Echocardiography assessment: Left ventricular ejection fraction (LVEF) ≥50%.
  6. 12-lead electrocardiogram evaluation: QTc<470ms.
* Female subjects should agree that contraceptive measures (such as intrauterine devices or condoms) must be used during the study period and within 6 months after the end of the study; the serum pregnancy test must be negative within 7 days before study enrollment, and must be Non-lactating subjects.

Exclusion Criteria:

* Tumor disease and medical history:

  1. Other malignant tumors that have occurred or are currently concurrently present within 3 years. The following conditions were eligible for enrollment: other malignancies treated with a single surgery, achieving 5 consecutive years of disease-free survival (DFS); cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta ( non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor-infiltrating basement membrane)];
  2. Pathologically suggested endometrial leiomyosarcoma, endometrial stromal sarcoma, undifferentiated uterine sarcoma or other high-grade sarcoma (Applicable to group 1 and 2), Pathologically suggested epithelial endometrial cancer or Carcinosarcoma (Applicable to group 3);
  3. The presence of tumor thrombus, spinal cord compression caused by bone metastases, brain metastases or cancerous meningitis;
  4. Imaging (CT or MRI) shows that the tumor has invaded around important blood vessels or the investigator judges that the tumor is very likely to invade important blood vessels and cause fatal bleeding during the follow-up study;
  5. Severe bone damage caused by tumor bone metastasis; including weight-bearing bone pathological fractures and spinal cord compression that occurred within 6 months or predicted by the investigator to be likely to occur in the near future;
  6. Uncontrolled pleural effusion, pericardial effusion or ascites judged by the investigator that still needs repeated drainage.
* Previous anti-tumor therapy or concomitant medication (the washout period is calculated from the end of the last treatment):

  1. Previously received anti-angiogenesis drugs, related immunotherapy drugs for PD-1, PD-L1, CTLA-4;
  2. Received drugs with immunomodulatory function, chemotherapy, radiotherapy, clinical trial drug treatment, traditional Chinese medicine or proprietary Chinese medicine with anti-tumor indications, or other anti-cancer therapy within 4 weeks before receiving the study drug for the first time;
  3. Received hormone therapy for endometrial cancer within 1 week before receiving the first study drug treatment;
  4. It is not satisfied that at least 5 half-lives have elapsed from the last use of the targeted drug to the first receiving of the study drug, if it is a combination drug, the drug with the longest half-life shall be calculated;
  5. Those who have undergone major surgery, major surgical treatment, incisional biopsy, obvious traumatic injury, or have not recovered sufficiently from previous surgery in the judgment of the investigator within 3 weeks before the first treatment with the study drug, or are expected to be required during the study period. Major surgery;
  6. The toxicity related to previous anti-tumor therapy has not recovered to CTCAE ≤ grade 1, except for alopecia and grade 2 peripheral neuropathy.
* Comorbid diseases and medical history:

  1. History of liver-related diseases: a. Decompensated cirrhosis; b. Active or chronic hepatitis; c. Bleeding disease secondary to hepatic insufficiency.
  2. Kidney related medical history: a. Renal failure requiring hemodialysis or peritoneal dialysis; b. Past or existing nephrotic syndrome, chronic nephritis.
  3. Cardiovascular and cerebrovascular related medical history: a. Suffering from epilepsy and requiring treatment; b. New York Heart Association class II-IV heart failure, second-degree or higher heart block, myocardial infarction within the past 6 months or Arterial thrombosis events, unstable arrhythmia or unstable angina; c. Cerebrovascular accident, cerebral infarction, etc. within 6 months; d. If the treatment can adequately control blood pressure, the group is allowed to enter the group; e. Past or current heart valve inflammation, endocarditis; f. Cardiovascular syncope, pathological ventricular arrhythmia.
  4. Gastrointestinal-related medical history: a. Inability to take oral medications; b. History of malabsorption syndrome or other diseases that interfere with gastrointestinal absorption; c. Active peptic ulcer or ulcerated lower gastrointestinal tract in the past 6 months Treated for inflammation; d. Persistent chronic diarrhea of grade 2 and above despite maximum medical treatment.
  5. Lung-related medical history: a. History of idiopathic pulmonary fibrosis, organized pneumonia, drug-induced pneumonia, idiopathic pneumonia, or evidence of active pneumonia found on chest CT scan during screening; b. Bronchodilator required Medically intervened bronchial asthma; c. The clinical manifestations are suspected to be tuberculosis, T-SPOT positive is judged by the investigator to have tuberculosis infection or active tuberculosis within 1 year before enrollment;
  6. Endocrine-related medical history: a. Poor control of type I or II diabetes; b. History of pituitary or adrenal dysfunction; c. Thyroid-stimulating hormone (TSH) > ULN, if T3 and T4 levels are normal, they can be enrolled.
  7. Immune-related medical history: a. A history of immunodeficiency, including HIV positive or other acquired and congenital immunodeficiency diseases; b. Organ transplantation planned or previously received, or hematopoietic stem cells received within 60 days before the first dose Transplant, or have obvious host transplant response; c. Active autoimmune disease; d. Systemic or topical immunosuppressive or hormonal therapy is required to achieve immunosuppression, and continue to be used within 7 days before the first dose Glucocorticoids, or patients who still need immunosuppressive drugs within 5 half-lives before the first dose.
  8. Bleeding risk: a. Suffering from bleeding (hemoptysis), coagulation disease or using warfarin, aspirin and other antiplatelet aggregation drugs (except aspirin ≤100 mg/d for prophylaxis); b. Regardless of severity, there are any signs or history of bleeding constitution; c. within 4 weeks before the first dose, any CTC AE ≥ grade 3 bleeding or bleeding events;
  9. The patient has an active systemic infection or an excessive viral load;
  10. Combining serious or not well-controlled diseases or diseases that the investigator determines may have a greater risk or affect the completion of the study, including but not limited to: a. History of clear neurological or mental disorders; b. Treponema pallidum specific antibody positive.
  11. Those who have a history of drug abuse and cannot quit or have a history of drug use.
* Research and treatment related:

  1. History of vaccination with live attenuated vaccine within 28 days before the start of study treatment, inactivated vaccine within 7 days, or planned vaccination during the study period;
  2. Those who have a history of severe allergic diseases, severe drug allergies, and are known to be allergic to macromolecular protein preparations or TQB2450 injection or any components in the prescription of Anlotinib capsules, their adjuvants and similar drugs;
* Subjects with insufficient compliance or other reasons are not suitable for enrollment after the investigator's assessment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Investigator-assessed objective response rate (ORR) | Through study completion, an average of 24 months
  The proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, including cases with complete remission and partial remission

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From data of randomization until the date of first documented progression or date death from any cause, whichever came first, assessed up to 24 months
  From randomization to the first occurrence of disease progression or death from any cause. Disease progression refers to tumor growth, or the metastasis of primary tumor lesions, or the discovery of new lesions, etc.
Overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 60 months
  From randomization to the time of death of death from any cause
Duration of Remission (DOR) | The length of time the patient received this regimen to keep the tumor shrinking, through study completion, an average of 24 months
  The period from the first judgment of complete remission (CR) or partial remission (PR) to the discovery of disease progression (PD).
Disease Control Rate (DCR) | Through study completion, an average of 24 months
  the proportion of patients whose tumors shrink or remain stable for a certain period of time, including complete remission (CR, Complete Response), partial remission (PR, Partial Response) and stable (SD, stable Disease) cases
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | Baseline to other antitumor therapy, through study completion, an average of 24 months
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).
Abnormal laboratory test indicators | Baseline to other antitumor therapy, through study completion, an average of 24 months
  The incidence of abnormal laboratory test indicators of participants by attachment 1 in the test protocol.
The surgical conversion rate | Baseline to other antitumor therapy, through study completion, an average of 24 months
  The proportion of subjects who meet the criteria and undergo radical resection surgery.

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - TianJin Medical University Cancer Institute & Hopspital, Tianjin, Tianjin Municipality